CLINICAL TRIAL: NCT00889837
Title: Pulmonary Safety of Staccato® Loxapine for Inhalation in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Staccato Loxapine Pulmonary Safety in Patients With COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMDC-004-108; 13 April 2009
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2009-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Staccato Loxapine; COPD; pulmonary safety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Inhaled Loxapine (Experimental): Staccato Loxapine, 10 mg doses x 2, 10 hours apart
  Interventions: Drug: Inhaled Loxapine
- Inhaled Placebo (Placebo Comparator): Staccato Placebo,inhalations x 2, 10 hours apart
  Interventions: Drug: Inhaled Placebo

INTERVENTIONS:
Drug: Inhaled Loxapine — Staccato Loxapine, 10 mg x 2 doses, 10 hours apart
  Arms: Inhaled Loxapine
Drug: Inhaled Placebo — Staccato Placebo, inhalations x 2 , 10 hours apart
  Arms: Inhaled Placebo

SUMMARY:
The purpose of this study is to assess the pulmonary safety of 2 doses of Staccato Loxapine within a day in patients with COPD.

DETAILED DESCRIPTION:
To address the possibility that inhalation of loxapine may have adverse pulmonary effects, we studied two 10-mg inhaled doses of loxapine or placebo were given 10 hr apart to subjects with chronic obstructive pulmonary disease (COPD). The objective was to determine the time course and reversibility of pulmonary effects for inhaled loxapine compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* History of COPD for at least 6 months with pre-bronchodilator FEV1 ≥40% of predicted value and >15 pack-year history of cigarette smoking.

Exclusion Criteria:

* History of asthma, or any other acute or chronic pulmonary disease.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 from baseline by spirometry | at each post-treatment time point (15 min to 34 hr)

SECONDARY OUTCOMES:
Change in FVC from baseline by spirometry | at each post-treatment time point (15 min to 34 hr)
Treatment emergent adverse events | Post-treatment time points

CONTACTS AND LOCATIONS:
Overall Officials: Mildred D. Gottwald, PharmD, Study Director — Alexza Pharmaceuticals, Inc.
Locations (1):
- Spartanburg Medical Research, Spartanburg, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Gross N, Greos LS, Meltzer EO, Spangenthal S, Fishman RS, Spyker DA, Cassella JV. Safety and tolerability of inhaled loxapine in subjects with asthma and chronic obstructive pulmonary disease--two randomized controlled trials. J Aerosol Med Pulm Drug Deliv. 2014 Dec;27(6):478-87. doi: 10.1089/jamp.2013.1114. PMID 24745666